CLINICAL TRIAL: NCT05951218
Title: Trigger Points of Supraspinatus Muscle: Osteopaths' Palpation Reproductibility and Ultrasound Translation
Brief Title: Effects of Inhibition Techniques Applied on Trigger Points of Supraspinatus Muscle on Echogenicity and Patients' Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut des Hautes Etudes Osteopathiques de Nantes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRIGGOSTEO-2; 2023-A00637-38 (Other: Agence nationale de sécurité du médicament et produits de santé)
Record Dates: First submitted 2023-07-09; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Pain
Keywords: trigger point; osteopathic palpation; ultrasound
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhibition technique (Experimental): In the first group, patients will receive inhibition treatment of the TP.
  Interventions: Other: inhibition technique
- placebo (Sham Comparator): The second group will receive a placebo treatment.
  Interventions: Other: placebo

INTERVENTIONS:
Other: inhibition technique — Inhibition treatment consists of applying progressive pressure with the finger until resistance is felt. The patient should feel discomfort but not pain. They should stop when they consider that the trigger point has been sufficiently relaxed. All the techniques should last less than 5 minutes. Osteopaths will be trained to have a close strength during techniques. The number of Newton that will be apply will be decided during training with the investigator
  Arms: inhibition technique
Other: placebo — The osteopath will perform a light touch on 4 areas for 30 seconds each time. The trigger point area must be lightly touched, followed by the upper part of the pectoralis major, the elbow and finally the anterior part of the opposite glenohumeral region.
  Osteopaths will be trained to have a close strength during techniques. The number of Newton that will be apply will be decided during training with the investigator with a palpatory pressure measurement tool. A proposition of 1N will be proposed to have a very light touch, without activating the C-tactile sensors.
  Arms: placebo

SUMMARY:
Trigger points (TP) are described as "hard, palpable nodules located within the taut bands of skeletal muscle".

The aim of this study is to evaluate the reproductibility of palpation of TP between osteopaths and to compare this perception to ultrasound measures of echogenicity.

Method:

A sample of 61 patients will be included in the study. An osteopath will determine the eligibility of the study. The supraclavicular area will be mark every 2 cm to establish a grid for all evaluations. All included osteopaths will receive a formation to test and treat with the same approach and the same strength during all stages.

First an osteopath will evaluate with palpation the presence of TP at every box of the grid.

A second osteopath will evaluate the same boxes and will be blinded to the result of the first osteopath.

At each step of palpation, a pain assessment will be carried out at each box. Then, the ultrasound technician will evaluate the echogenicity of every box and will be blinded to the prior results.

Every patient with a TP diagnosed by the first osteopath, will be randomised into two groups (inhibition of trigger point technique with a long standing press on the TP, placebo technique with four light touch techniques on both shoulders, sternum and rachis).

The second osteopath will evaluate the same boxes and will be blinded to the randomisation process. At each step of palpation, a pain assessment will be carried out at each box.

The ultrasound technician will evaluate an other time the echogenicity of every box and will be blinded to the prior results, and randomisation.

A blinded statistician will evaluate the efficacy of inhibition technique on echogenicity and patients' pain during the tests.

The protocol has been approved by a french ethic committee.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years
* be affiliated to a social security system or benefit from such a system.

Exclusion Criteria:

* pregnant or breast-feeding women
* adults under guardianship
* patients under protection
* history of tegumentary or muscular damage in the area concerned
* wish to stop the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-08-29 (Estimated); Primary Completion 2024-08-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain during palpation at 5 minutes | 5 minutes before and 5 minutes after the treatment session
  change in pain will be assess with a 0 to 4 scale before and after techniques on each boxes. Pain in relation to a TP will be compared between patients from placebo arm and intervention arm

SECONDARY OUTCOMES:
Change from baseline echogenicity at 5 minutes | 5 minutes before and 5 minutes after the treatment session
  Echogenicity will be assess with a binary outcome (0 for normal echogenicity and 1 for hypoechogenicity) before and after techniques on each boxes. Echogenicity in relation to a TP will be compared between patients from placebo arm and intervention arm

IPD SHARING:
Plan to Share IPD: Yes
on demand to M. Salmon
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code